CLINICAL TRIAL: NCT03363126
Title: Visual Outcome After Transsphenoidal Surgery for Pituitary Macroadenoma
Acronym: RetroADEN
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20160404_1_WEI
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Pituitary Tumor; Optic Chiasm Disorder
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endonasal transsphenoidal pituitary tumor removal — Removal of pituitary tumor by transsphenoidal endonasal surgery

SUMMARY:
Endoscopic endonasal transsphenoidal surgery is a procedure for the treatment of pituitary macroadenomas that cause visual impairment through optic chiasm compression. The aim of this retrospective study is to describe visual outcome after this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pituitary tumor causing optic chiasm compression (documented on MRI or CT-scan)
* Visual impairment caused by chiasm compression
* Treatment by transsphenoidal endonasal surgery
* Treatment in the Rothschild Foundation (Paris) between 2009 and 2013

Exclusion Criteria:

* Ophtalmologic condition other than optic chiasm compression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the Rothschild Foundation (Paris) between 2009 and 2013 by transsphenoidal endonasal surgery for pituitary tumor causing optic chiasm compression and visual disorders
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Post-operative gain in visual acuity | six months
  Difference between pre-operative and post-operative visual acuity, expressed in LogMAR

IPD SHARING:
Plan to Share IPD: No